CLINICAL TRIAL: NCT02184650
Title: Early Nutrition and Neurological Development of Very Preterm Infants
Brief Title: Nutrition and Neurological Development of Very Preterm Infants
Acronym: EPINUTRI_3
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 13016; ID RCB 2014-A00941-46 (Other: France: Ministry of Health)
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Premature Infant; Infant Nutrition Disorders; Delayed Mental Development
Keywords: Premature infants; Nutritional status; Polyunsaturated fatty acids status
MeSH Terms: conditions — Premature Birth; Infant Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — saliva, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Premature infants: Premature infants with a GA < 32 weeks
  Interventions: Other: Premature infants with a GA < 32 weeks

INTERVENTIONS:
Other: Premature infants with a GA < 32 weeks — At 3 years of age: ASQ (filled in by parents)

SUMMARY:
The main goal of this study is to determine, in preterm infants born with a GA < 32 weeks, the association between:

* the quantity of mother's milk and duration and breastfeeding
* the intake of polyunsaturated fatty acids and iron during hospitalizations

DETAILED DESCRIPTION:
The main hypothesis of this study is that the intake of lipid during hospitalization in neonatology department is associated with neurological development of preterm infants born with a GA < 32 weeks. The other hypotheses are that iron intake and the duration of breastfeeding are also associated with the development of preterm infants.

In the previous study EPINUTRI (NCT01486173), the development of infants was evaluated until the age of 1 year. EPINUTRI_3 is the follow-up of EPINUTRI until the age of 3 years.

The aim of EPINUTRI_3 study is to determine the association between lipid intake during hospitalization in neonatology department of preterm infants born with a GA < 32 weeks.

The secondary objective is :

- to evaluate the association between these factors and communication, developmental and social-emotional delays with the test " Ages and Stages questionnaire " (ASQ) at 3 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants previously included in EPINUTRI study
* Non opposition of the parents for the collection of clinical and nutritional data

Exclusion Criteria:

* Refusal of the parents to collect clinical and nutritional data

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subsample of infants born very preterm (before 32 weeks of gestation), otherwise included in the French national cohort EPIPAGE 2, and previously included in EPINUTRI study.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Neurological development | At 3 years of age
  Age and Stages Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lapillonne, M.D, Ph.D., Principal Investigator — Hôpital Necker Assistance Publique-Hôpitaux de Paris
Locations (1):
- Hôpital Necker Assistance Publique- Hôpitaux de Paris, Paris, France

REFERENCES:
- [Result] Pierrat V, Marchand-Martin L, Marret S, Arnaud C, Benhammou V, Cambonie G, Debillon T, Dufourg MN, Gire C, Goffinet F, Kaminski M, Lapillonne A, Morgan AS, Roze JC, Twilhaar S, Charles MA, Ancel PY; EPIPAGE-2 writing group. Neurodevelopmental outcomes at age 5 among children born preterm: EPIPAGE-2 cohort study. BMJ. 2021 Apr 28;373:n741. doi: 10.1136/bmj.n741. PMID 33910920